CLINICAL TRIAL: NCT05701436
Title: Applicability of 3D Histoculture Drug Response Assay(3D-HDRA) in Patients With Primary Liver Cancer: A Randomized Controlled Trial
Brief Title: Applicability of 3D-HDRA in Patients With Primary Liver Cancer: A Randomized Controlled Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-KY-277-01
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-01

CONDITIONS: Liver, Cancer of, Primary Resectable
MeSH Terms: interventions — Oxaliplatin; Doxorubicin; lobaplatin; Cisplatin; Leucovorin; Fluorouracil; raltitrexed

STUDY DESIGN:
Intervention Model Description: The test group received postoperative conventional treatment combined with precise transarterial chemoembolization based on 3D-HDRA results, and the control group received postoperative conventional treatment combined with Empirical transarterial chemoembolization.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- the test group (Experimental): The test group received postoperative conventional treatment combined with precise transarterial chemoembolization based on 3D-HDRA results. Precise transarterial chemoembolization at 1-month intervals for 4 months after surgery.
  Interventions: Drug: Oxaliplatin; Drug: Doxorubicin; Drug: Lobaplatin; Drug: Cisplatin; Drug: Oxaliplatin, Leucovorin, fluorouracil; Drug: Lobaplatin, Raltitrexed
- the control group (Active Comparator): The control group received postoperative conventional treatment combined with Empirical transarterial chemoembolization. Empirical transarterial chemoembolization at 1-month intervals for 4 months after surgery.
  Interventions: Drug: Oxaliplatin; Drug: Doxorubicin; Drug: Lobaplatin; Drug: Cisplatin; Drug: Oxaliplatin, Leucovorin, fluorouracil; Drug: Lobaplatin, Raltitrexed

INTERVENTIONS:
Drug: Oxaliplatin — 130 mg per square body surface area for a total of four transcatheter hepatic artery infusions per month.
Drug: Doxorubicin — 20 mg per square body surface area for a total of four transcatheter hepatic artery infusions per month.
Drug: Lobaplatin — 50 mg per square body surface area for a total of four transcatheter hepatic artery infusions per month.
Drug: Cisplatin — 50 mg per square body surface area was used for monthly transhepatic arterial infusions.
Drug: Oxaliplatin, Leucovorin, fluorouracil — Oxaliplatin(130 mg per square body surface area), Leucovorin(400 mg per square body surface area), and fluorouracil(2800 mg per square body surface area) were used for monthly transhepatic arterial infusions.
Drug: Lobaplatin, Raltitrexed — Lobaplatin(50 mg per square body surface area) and Raltitrexed(3 mg per square body surface area) were used for monthly transhepatic arterial infusions.

SUMMARY:
This Randomized Controlled Trial was to clarity the clinical feasibility of 3D-HDRA results in guiding the drug use of interventional chemotherapy after primary liver cancer surgery.

DETAILED DESCRIPTION:
Data of Patients who received 3D-HDRA after primary liver cancer radical reaction and received Transarterial Chemoembolization #will be collected #excluding incomplete data.

The primary endpoint was the one-year disease-free survival(DFS) rate #Secondary endpoint was the adverse event.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily cooperated with the study and signed an informed consent form.
2. Any gender, age 18 or older, 75 or younger.
3. Patients who need to confirm the maximum tumor load (the maximum diameter of a single tumor lesion) before performing radical surgery; patients with a confirmed diagnosis of primary liver cancer after postoperative pathological histological examination.
4. Patients with R0 resection confirmed by imaging and pathology (no residual lesions and complete tumor resection after radical surgery).
5. Child-Pugh score of 5-7 (A or B), patients with a score of 7 must be free of ascites.
6. ECOG physical fitness status score of 0-1.
7. Women of childbearing age with a negative pregnancy test and willing to use effective contraception for the duration of the study.

Exclusion Criteria:

1. Patients with recurrent liver cancer.
2. Patients with existing extrahepatic distant metastases (including local lymph node metastases or distant organ metastases: e.g., lung, brain, bone, etc.) at the time of diagnosis.
3. Treatment with other experimental drugs or other interventions after radical resection.
4. Patients with other malignant tumors that have not been cured within 5 years.
5. Patients with non-radical resections (R1 and R2 resections).
6. Patients with residual or recurrent lesions detected on imaging within 1-2 months after surgery.
7. Patients in whom death occurred within 30 days after surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
The one-year DFS rate | From the start date of the Treatment until date of the time of 1 year
  The one-year DFS rate is defined as the percentage of participants who have not accrued disease at the time of 1 year

SECONDARY OUTCOMES:
Adverse events | From the beginning of therapy until the date of death from any cause(max 24 months)
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Mingxin Pan, Prof, Study Director — Study Principal Investigator Southern Medical University, China
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China